CLINICAL TRIAL: NCT00151151
Title: The S.A.F.E. Study: Computer-Aided Counseling to Prevent Teen Pregnancy/STDs - Validity and Reliability Testing of Computer Measures, Pilot-testing of Timeline Followback Calendar Protocol, and Randomized Efficacy Study
Brief Title: The S.A.F.E. Study : Computer-Aided Counseling to Prevent Teen Pregnancy/Sexually Transmitted Diseases (STDs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0405473; HD41058
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2008-01

CONDITIONS: Pregnancy; Sexually Transmitted Diseases
Keywords: pregnancy prevention; STD prevention; adolescents; motivational interviewing; abstinence; contraception; transtheoretical model; sexual behavior
MeSH Terms: conditions — Sexually Transmitted Diseases; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Computer-Assisted Motivational Intervention
Behavioral: Didactic Educational Counseling

SUMMARY:
This is a randomized clinical trial assessing the efficacy of two types of counseling (Computer-Assisted Motivational Intervention [CAMI] versus Didactic Educational Counseling [DEC]) to see which can better reduce female adolescents' risk taking behaviors that put them at risk for unintended pregnancy and sexually transmitted diseases (STDs). The intervention phase consists of three 30-minute counseling sessions over the first 6 months followed by a visit every three months during the 12 month follow up phase. We, the researchers, hypothesize that the CAMI will decrease the proportion of subjects who engage in any intercourse that is poorly protected against pregnancy and against STDs.

DETAILED DESCRIPTION:
Adolescent unintended pregnancy and STDs remain at epidemic levels in the United States. Healthy People 2010 Objectives set a goal to increase to 90% the proportion of sexually active adolescents who use contraception that both effectively prevents pregnancy and provides barrier protection against disease. How to effectively counsel adolescents to reach this goal is unclear. Counseling and feedback based on the Transtheoretical Model (TTM) have demonstrated greater success than standard, action-oriented advice in several domains of behavior change. The effectiveness of this type of counseling to alter female adolescents' sexual and contraceptive behaviors has not been rigorously evaluated. We propose recruiting 660 female adolescents, ages 13 to 21 years, from an inner-city, hospital-based clinic and randomizing them to either an innovative Computer-Assisted Motivational Intervention (CAMI) or a Didactic Educational Control (DEC). The CAMI group will receive three, 30-minute sessions of one-on-one counseling with a counselor that is guided by computer-generated personalized feedback. The CAMI is based on the principles of the TTM and on Motivational Interviewing. The DEC provides three 30-minute sessions of one-on-one didactic information on contraception, STD prevention, and abstinence. The two interventions are identical in length and timing but vary in educational content, counseling style, and the provision of personalized feedback. We will track the two groups of female adolescents in this study through a 6-month intervention phase and a 12-month follow-up phase to assess differences in sexual and contraceptive behaviors by group. The primary specific aim for the study is to evaluate the efficacy of the CAMI as compared to the DEC in reducing sexual behaviors that increase the risks of both unintended pregnancy and STDs. We will examine protective sexual behaviors in three ways: 1) behaviors that protect against pregnancy; 2) behaviors that protect against STDs; and 3) behaviors that protect against both pregnancy and STDs. Our primary hypothesis is that the CAMI will decrease the proportion of subjects who engage in any intercourse that is poorly protected against pregnancy and against STDs. We also predict that among sexually active subjects, the CAMI will increase the percentage of episodes of intercourse that are well protected by the use of both condoms plus another contraceptive. Finally, we also predict that the CAMI will increase the prevalence of abstinence among the entire sample. If proven effective, computer-assisted personalized motivational counseling could be broadly implemented as a method to decrease the incidence of unintended pregnancy and STDs among female adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescents,
* Ages 13 to 21 years of age,
* Not currently pregnant or planning pregnancy in next 18 months,
* English speaking,
* Able to return every 3 months to study office for 18 months

Exclusion Criteria:

* Medically or surgically sterile,
* Has intrauterine device (IUD) or subdermal contraceptive implant,
* Hearing or visual impairments that might interfere with using the computerized assessment or participating in counseling session,
* In foster care or on house arrest,
* Has sex exclusively with female partners

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 660 (Estimated)
Dates: Start 2003-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Self-reported sexual and contraceptive behaviors recorded by a 90-day timeline follow back interview at 9 and 18 months compared to baseline

SECONDARY OUTCOMES:
Stage of readiness to be abstinent, use condoms, spermicide, and hormonal contraception based on a computerized assessment
Reported drug and alcohol use recorded by a 90-day timeline follow back interview

CONTACTS AND LOCATIONS:
Overall Officials: Melanie A. Gold, DO, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States